CLINICAL TRIAL: NCT03320629
Title: A Prospective Study of Apatinib Plus Radiotherapy and S-1 for Treatment of Refractory or Metastatic Esophageal Squamous Cell Carcinoma
Brief Title: A Study of Apatinib Plus Radiotherapy and S-1 for Treatment of Refractory or Metastatic Esophageal Squamous Cell Carcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: This study was voluntarily terminated after investigator assessment, with no safety concerns identified related to the trial intervention or procedures. The primary reason for termination was difficulty in patient recruitment.
Sponsor: Hebei Medical University Fourth Hospital (Other)
Responsible Party: Principal Investigator, Jun wang, Director of radiotherapy department1, Hebei Medical University Fourth Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HRA-E01
Record Dates: First submitted 2017-10-20; First posted 2017-10-25 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2017-10

CONDITIONS: Refractory or Metastatic Esophageal Squamous Cell Carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- apatinib and S-1 radiotherapy (Experimental): apatinib 500mg qd po S-1 40-60mg/time bid po d1-14 q3w radiotherapy 50-60Gy/25-30times until disease progression or intolerable toxicity or patients withdrawal of consent
  Interventions: Combination Product: apatinib S-1 radiotherapy
- S-1 radiotherapy (Active Comparator): S-1 40-60mg/time bid po d1-14 q3w radiotherapy 50-60Gy/25-30times until disease progression or intolerable toxicity or patients withdrawal of consent
  Interventions: Combination Product: S-1 radiotherapy

INTERVENTIONS:
Combination Product: apatinib S-1 radiotherapy — apatinib 500mg qd po S-1 40-60mg/time bid po d1-14 q3w radiotherapy 50-60Gy/25-30times until disease progression or intolerable toxicity or patients withdrawal of consent
  Arms: apatinib and S-1 radiotherapy
Combination Product: S-1 radiotherapy — S-1 40-60mg/time bid po d1-14 q3w radiotherapy 50-60Gy/25-30times until disease progression or intolerable toxicity or patients withdrawal of consent
  Arms: S-1 radiotherapy

SUMMARY:
The purpose of this study is to assess the efficacy and safety of patients who receive apatinib plus radiotherapy and S-1 for treatment of refractory or metastatic esophageal squamous cell carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age:18 to 70 years old (man or female); 2. Imageology diagnosed with refractory or metastatic esophageal squamous cell carcinoma(pathologically diagnosed with supraclavicular lymph node metastasis and anastomotic recurrence ); 3. The distant metastatic is oligotransfera, with radiotherapy indication; 4. Patients with measurable lesions(measuring≥10mm on spiral CT scan, satisfying the criteria in RECIST1.1); 5. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2; 6. Major organ function has to meet the following certeria:

  1. For results of blood routine test (without blood transfusion within 14 days)

     1. HB≥100g/L;
     2. ANC≥3.0×109/L;
     3. PLT≥100×109/L;
  2. For results of blood biochemical test：

     1. TBIL<1.5×ULN；
     2. ALT and AST<2.5×ULN, but< 5×ULN if the transferanse elevation is due to liver metastases；
     3. Serum creatinine ≤1ULN , calculated creatinine clearance>50 ml/min(per the Cockcroft-Gault formula); 7. Life expectancy greater than or equal to 3 months; 8. Women of childbearing age must have contraceptive measures or have test pregnancy (serum or urine) enroll the study before 7 days, and the results must be negative, and take the methods of contraception during the test and the last to have drugs after 8 weeks. Men must be contraception or has sterilization surgery during the test and the last to have drugs after 8 weeks; 9. Coagulation function is normal, without active hemorrhage and thrombosis:

     <!-- -->

     1. INR<1.5×ULN
     2. APTT<1.5×ULN
     3. PT<1.5ULN 10. Participants were willing to join in this study, and written informed consent; 11. Participants were good adherence, cooperate with the follow-up.

Exclusion Criteria:

* 1. Allergic to apatinib; 2. Have high blood pressure and antihypertensive drug treatment can not control (systolic blood pressure > 140 mmHg, diastolic blood pressure > 90 mmHg), with classⅡand above coronary heart disease and arrhythmia (including QTc lengthened men > 450 ms, women > 470 ms) and cardiac insufficiency; 3. A variety of factors influencing oral drugs (such as unable to swallow, nausea, vomiting, chronic diarrhea and intestinal obstruction, etc.); 4. Patients with tendency of gastrointestinal bleeding, including the following;

  1. Active ulcerative lesions, and defecate occult blood (+ +);
  2. Has melena and hematemesis in three months;
  3. For defecate occult blood (+) or(+/-) ,must be received gastroscopy, the physicians consider there are potential bleeding risk with ulcers, hemorrhagic diseases; 5. Coagulant function abnormality (INR > 1.5 ULN, APTT > 1.5 ULN), with bleeding tendency; 6. Patients with thrombosis or anticoagulant drug therapy; 7. Patients with symptoms of central nervous system metastasis; Patients with other malignant tumors within 5 years (except for the treated skin basal cell carcinoma and cervical carcinoma in situ); 8. history of psychiatric drugs abuse and can't quit or patients with mental disorders; 9. Less than 4 weeks from the last clinical trial; 10. Have received prior treatment with anti- VEGF/VEGFR; 11. Researchers considered there are serious harm to patient safety or affect the patients who have completed the study; 12. Pregnant or lactating women; 13. The researchers think inappropriate.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2017-11-01 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Progression free survival | evaluated in 24 months since the treatment began
  Baseline to measured date of progression or death from any cause

SECONDARY OUTCOMES:
Overall survival | the first day of treatment to death or last survival confirm date，up to 24 months
  Baseline to measured date of death from any cause
Disease control rate | tumor assessment every 6 weeks ，up to 24 month
  Baseline to measured progressive disease
Objective response rate | tumor assessment every 6 weeks，up to 24 months
  Baseline to measured stable disease
Side effects | evaluated in the 24th month since the treatment began according to the Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0
  throughout study

CONTACTS AND LOCATIONS:
Locations (1):
- Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei, China